CLINICAL TRIAL: NCT04123054
Title: An Open-Label, Randomized, Two-Way, Parallel Study to Compare the Effectiveness of Multiple Daily Injection Treatment With an Insulin Dose Optimization Algorithm in Free-Living Outpatient Conditions in Patients With Type 1 Diabetes
Brief Title: A Novel mHealth Application Guided by an Optimization Algorithm for T1D Sensor-Augmented Insulin Injection Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-5887
Record Dates: First submitted 2019-08-15; First posted 2019-10-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1
Keywords: Multiple Daily Injections,; Type 1 diabetes; Optimization algorithm
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, controlled, two-way parallel study to compare glucose control between sensor-augmented MDI therapy and our basal-bolus optimizing algorithm over 3 months. Adults with type 1 diabetes who are enrolled in the study will randomly undergo one of the two interventions for the entire study duration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensor-Augmented MDI + Mobile App (control) (Active Comparator): Participants will continue their usual multiple daily injections (MDI) therapy along with the use of Freestyle Libre glucose sensors (Abbott Diabetes Care) and a mobile application that facilitates insulin dose calculations while collecting insulin and meal data.
  Interventions: Device: Mobile App
- Sensor-Augmented MDI + Mobile App + Basal-Bolus Optimization Algorithm (Experimental): Participants will undergo multiple daily injections (MDI) therapy along with the use of Freestyle Libre glucose sensors (Abbott Diabetes Care) and a mobile application that facilitates insulin dose calculations while collecting insulin and meal data. Every week, participants' insulin doses will be updated by the optimization algorithm's recommendations.
  Interventions: Device: Mobile App + Basal-Bolus Optimization Algorithm

INTERVENTIONS:
Device: Mobile App — Participants will use the mobile app to log their daily basal dose and calculate their meal doses by entering their sensor glucose value (and amount of meal carbohydrates if applicable) using the built-in bolus calculator.
  Arms: Sensor-Augmented MDI + Mobile App (control)
Device: Mobile App + Basal-Bolus Optimization Algorithm — Participants will use the mobile app to log their daily basal dose and calculate their meal doses by entering their sensor glucose value (and amount of meal carbohydrates if applicable) using the built-in bolus calculator. In addition, participants will receive weekly app notifications with personalized recommendations for insulin parameter adjustments made by the optimization algorithm.
  Arms: Sensor-Augmented MDI + Mobile App + Basal-Bolus Optimization Algorithm

SUMMARY:
The Artificial Pancreas lab at McGill University has developed an optimization algorithm for adults with Type 1 Diabetes (T1D) on Multiple Daily Injection (MDI) therapy with the adjunctive use of glucose sensor technology, collectively known as sensor-augmented MDI therapy. The algorithm is designed to estimate optimal basal-bolus parameters based on the patient's glucose, insulin and meal data over several days. The investigators hope that this algorithm will be better able to improve long-term glycemic targets by reducing HbA1c levels compared to sensor-augmented MDI therapy alone.

DETAILED DESCRIPTION:
The changes in eligibility criteria indicated below are from a previously approved amendment but were inadvertently omitted in the previous PRS update made in November of 2020. Therefore, this note serves to clarify the order of updates.

Inclusion: HbA1c ≥ 7.5% in the last 2 months (modification)

Exclusion:

* More than 1 slow-acting injection and unwilling to switch to once a day for the study (addition)
* Severe hypoglycemic episode within one month of admission (addition)

In the subsequent amendment, we modified the timeframe for the HbA1c inclusion criterion to obtain a more accurate representation of their current glucose control at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age
2. Clinical diagnosis of type 1 diabetes for at least 12 months. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
3. Undergoing multiple daily injection therapy.
4. Baseline HbA1c value ≥ 7.5% (up to 7 days before or after screening).

Exclusion Criteria:

1. Serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
2. Failure to comply with the study protocol or with the team's recommendations.
3. Injection of isophane insulin (NPH) or any intermediate-acting insulin
4. More than 1 slow-acting injection and unwilling to switch to once a day for the study
5. Current or ≤ 1-month use of other antihyperglycemic agents (Sodium-Glucose Cotransporter 2 inhibitor (SGLT2), Glucagon-Like Peptide-1 (GLP-1), Metformin, Acarbose, etc.…).
6. Pregnancy
7. Severe hypoglycemic episode within one month of admission.
8. Severe diabetic ketoacidosis episode within one month of admission
9. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator
10. Recent (<6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery
11. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels | Pre-intervention and post-intervention, approximately 12 weeks
  Difference in HbA1c levels from the start to the end of the study

SECONDARY OUTCOMES:
The number of patients that achieve an HbA1c at the end-of-study visit of: | Post-intervention, approximately 12 weeks
  a. less than or equal to 7.0%; b. less than or equal to 6.5%
Percentage of time of sensor glucose levels spent: | 12 weeks
  a. between 3.9 and 7.8 mmol/L; b.between 3.9 and 10 mmol/L; c. below 3.9 mmol/L; d.below 3.3 mmol/L; e.below 2.8 mmol/L; f. above 7.8 mmol/L; g. above 10 mmol/L; h. above 13.9 mmol/L; i. above 16.7 mmol/L.
Percentage of overnight time (23:00-7:00) of sensor glucose levels: | 12 weeks
  a. between 3.9 and 7.8 mmol/L; b. between 3.9 and 10 mmol/L; c.below 3.9 mmol/L; d. below 3.3 mmol/L; e. below 2.8 mmol/L; f. above 7.8 mmol/L; g. above 10 mmol/L; h. above 13.9 mmol/L; i. above 16.7 mmol/L.
Percentage of daytime (7:00-23:00) of sensor glucose levels: | 12 weeks
  a. between 3.9 and 7.8 mmol/L; b. between 3.9 and 10 mmol/L; c. below 3.9 mmol/L; d. below 3.3 mmol/L; e. below 2.8 mmol/L; f. above 7.8 mmol/L; g. above 10 mmol/L; h. above 13.9 mmol/L; i. above 16.7 mmol/L.
Standard deviation of glucose levels. | 12 weeks
  Standard deviation of glucose levels as a measure of glucose variability.
Total insulin delivery. | 12 weeks
  Total insulin delivery
Mean sensor glucose level during: | 12 weeks
  a. the overall study period; b. the daytime period; c. overnight period.

OTHER OUTCOMES:
Mean scores of the survey items on modified versions of the Diabetes Treatment Satisfaction Questionnaire | Pre-intervention, then monthly, approximately 12 weeks
  Scoring for treatment satisfaction ranges from 0-6; higher score = higher satisfaction (patient-reported outcomes)
Mean scores of the survey items on modified versions of the Mobile Health App Usability Questionnaire | Post-intervention, approximately 12 weeks
  Scoring for the usability of the app ranges from 1-7; higher score = higher usability (patient-reported outcomes)
Recurrent themes from semi-structured interviews | Post-intervention, approximately 12 weeks
  Qualitative interview data to obtain an understanding of relationships by connecting lived experiences with a) mean survey scores and b) primary and secondary outcomes regarding the use of the study software on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tsoukas, MD, Principal Investigator — RI-MUHC
Locations (2):
- Canada (2):
  - CIUSSS West-Central Montreal, Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Participant data - after de-identification.
Supporting Information: Study Protocol
Time Frame: Within one year of publication.
Access Criteria: Access provided upon reasonable request.

REFERENCES:
- [Derived] Kobayati A, El Fathi A, Garfield N, Legault L, Jafar A, Yale JF, Tsoukas MA, Haidar A. A Bayesian decision support system for automated insulin doses in adults with type 1 diabetes on multiple daily injections: a randomized controlled trial. Nat Commun. 2025 Sep 29;16(1):8593. doi: 10.1038/s41467-025-63671-0. PMID 41022835